CLINICAL TRIAL: NCT00669708
Title: kühlender Effekt Der Eucerin pH5 Lotion Und Der Eucerin pH5 Lotion Mit Cooling Compound Bei Trockener, Juckender Haut
Brief Title: Topical Therapy With Cooling Effect in Dry Itchy Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Prof. Dr. Sonja Ständer, Department of Dermatology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SST-Pr-12-2007; 2007-510-f-S
Record Dates: First submitted 2008-04-22; First posted 2008-04-30 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-02

CONDITIONS: Compensate the Roughness of the Skin; Compensate the Sensory Symptoms
Keywords: dry skin; cooling; itch
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): ph5 Eucerin Lotion with cooling compound
  Interventions: Device: cooling compound (ph5 Eucerin)
- 2 (Placebo Comparator): ph5 Eucerin Lotion
  Interventions: Device: cooling compound (ph5 Eucerin)

INTERVENTIONS:
Device: cooling compound (ph5 Eucerin) — application twice daily to the skin
  Other Names: ph5 Eucerin

SUMMARY:
Dry skin is a physiological condition and is characterized in contrast to greasy skin by roughness, desquamation and lack of brightness of the skin surface. Subjectively, feelings of tension, burning and itching can occur. The skin reacts more intensive on external and physical noxae. Dry skin is caused by a lack of moisture. This is most common during the winter months, when heating systems dry the air. Bathing with hot water, spending extended periods of time in the hot sun, and the skin's natural aging process also remove moisture and oils from the skin. It is diagnosed through clinical observation. People suffering from dry skin often desire to improve this condition for optical cosmetic reasons and due to the occasional feeling of tension. The aim of this investigation is to observe the improvement (or not) of dry itchy skin by a lotion containing a cooling compound

DETAILED DESCRIPTION:
The patient use the lotion twice daily for a four-week period. Additionally, the patient receives a documentation sheets to note several parameters. In a sensory assessment, product specific parameter such as spreadability, permeability, lubricating, smell of lotion and cosmetic acceptance during the treatment will be assessed (at the beginning, after 2 weeks, after 4 weeks, 2 weeks after stopping treatment). Before and after skin care measurement, the skin surface will be investigated by d-squames and corneometer. After four weeks the skin care measurement will be terminated and the patient can continue with a treatment of his choice. A monitoring of at least 70 patients is intended.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age: over 18 years
2. itch over VAS 3

Exclusion Criteria:

1. pregnancy, lactating women
2. drug abuse
3. active psychosomatic and psychiatric disease
4. active cancer.
5. topical application of tacrolimus, pimecrolimus, corticosteroids or capsaicin two weeks before study start
6. intake of antihistamines, corticosteroids, cyclosporine A and other immunosuppressants, naltrexone, UV-therapy two weeks before study start
7. participation in any other research study during the previous 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Compensate the roughness of the skin Compensate sensory symptoms | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Ständer, MD, Principal Investigator — Department of Dermatology, University of Münster
Locations (1):
- Department of Dermatology, University of Münster, Münster, Germany

REFERENCES:
- [Derived] Stander S, Augustin M, Roggenkamp D, Blome C, Heitkemper T, Worthmann AC, Neufang G. Novel TRPM8 agonist cooling compound against chronic itch: results from a randomized, double-blind, controlled, pilot study in dry skin. J Eur Acad Dermatol Venereol. 2017 Jun;31(6):1064-1068. doi: 10.1111/jdv.14041. Epub 2016 Dec 7. PMID 27862339